CLINICAL TRIAL: NCT03531957
Title: A Randomized, Double-blind, Placebo-controlled, Phase 2B Study to Evaluate the Efficacy, Safety, Tolerability, and Pharmacokinetics of ASN002 in Subjects With Moderate to Severe Atopic Dermatitis
Brief Title: Phase 2B Study to Evaluate ASN002 in Subjects With Moderate to Severe Atopic Dermatitis (RADIANT)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Asana BioSciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ASN002AD-201
Record Dates: First submitted 2018-04-19; First posted 2018-05-22 (Actual); Results first posted 2022-11-15 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Atopic Dermatitis
Keywords: eczema
MeSH Terms: conditions — Dermatitis, Atopic; Eczema | interventions — gusacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- ASN002 40 mg (Experimental): 40 mg ASN002
  Interventions: Drug: ASN002
- ASN002 60 mg (Experimental): 60 mg ASN002
  Interventions: Drug: ASN002
- ASN002 80 mg (Experimental): 80 mg ASN002
  Interventions: Drug: ASN002
- Placebo Oral Tablet (Experimental): Matching placebo for ASN002 doses
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: ASN002 — Daily dose of ASN002 for 12 weeks
  Arms: ASN002 40 mg; ASN002 60 mg; ASN002 80 mg
Drug: Placebo Oral Tablet — Placebo of ASN002 for 12 weeks
  Arms: Placebo Oral Tablet

SUMMARY:
This is a randomized double-blind/placebo study evaluate the efficacy of ASN002 in subjects with moderate to severe atopic dermatitis (AD).

DETAILED DESCRIPTION:
This is a placebo controlled study where subjects with moderate to severe atopic dermatitis will be randomized (1:1:1:1) to receive ASN002 at 40 mg, 60 mg, or 80 mg, or placebo once daily for 12 weeks. Eligible subjects will get the opportunity to enroll in the 24 month open-label extension study (OLE). There will be a 4-week follow up period for subjects not participating in the OLE study. This study will also characterize the pharmacokinetics and pharmacodynamics of ASN002 through blood sampling and three or four biopsies from subjects who consent.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained prior to any study-related procedure being performed;

  * Male or female, 18≤ years and ≤75 years of age with chronic AD for at least 6 months.
  * At least 10% body surface area (BSA) of AD involvement at the baseline visits
  * Has a body mass index (BMI) ≤35 kg/m2
  * History of inadequate response to topical corticosteroids or calcineurin inhibitors as treatment for AD within 1 year before the screening visit.
  * Willing to apply only a basic bland emollient once or twice-daily for at least 7 days before the baseline visit.
  * Willing to comply with discontinuation of certain treatments for AD, as directed by the Investigator.
  * Willing to use medically effective methods of birth control
  * Females of reproductive potential must have a negative serum pregnancy test at screening and negative urine pregnancy test at Day 1..
  * Willing and able to comply with clinic visits and study-related procedures

Exclusion Criteria:

* Clinically infected atopic dermatitis.

  * Presence of any of the following laboratory abnormalities at the screening visit: Hemoglobin < 11 g/dL, White blood cell (WBC) < 3.0 x 103 /μL, Platelet count < 125 x 103 /μL, Neutrophils < < 2.50 x 103 /μL, Lymphocytes ≤ 1.2 x 103 /μL, Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) > 1.5 x the upper limit of normal (ULN),Total bilirubin > ULN (except for elevated indirect bilirubin secondary to Gilbert's syndrome), Creatinine > ULN
  * A serious uncontrolled condition including hypertension, history of tuberculosis, hepatitis B or C infection, immune deficiency, heart disease, heart conduction disorder, diverticulitis, diabetes, reflux disease requiring protocol pump inhibitor therapy, malabsorption syndrome, or cancer.
  * Any condition requiring the use of anticoagulants.
  * History of hypertrophic scarring or keloid formation in scars or suture sites.
  * Any medical or psychiatric condition which, in the opinion of the investigator or the sponsor's medical monitor, would place the patient at risk, interfere with participation in the study, or interfere with the interpretation of study results
  * Pregnant or breast-feeding women
  * Known hypersensitivity to ASN002 or its excipients;
  * Prior treatment with SYK or JAK inhibitors for which the subject received no clinical benefit, or the subject relapsed whilst on therapy.
  * Has received any marketed or investigational biological agent within 12 weeks or 5 half-lives (whichever is longer) prior to Day 1.
  * Planned major surgical procedure during the length of the patient's participation in this study
  * There will be a waiting period of 4 weeks before receiving the first does for anyone who has used oral or intravenous treatments (other than biologics) that could affect atopic dermatitis, received a non-biological investigational product or device, excessive sun exposure, is planning a trip to a sunny climate, or has used tanning booths, or received or plans to receive a live attenuated vaccine one four weeks after the last day of taking the drug.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Actual)
Dates: Start 2018-07-05 (Actual); Primary Completion 2019-07-22 (Actual); Study Completion 2019-08-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Zammit, Ph.D., Study Director — Asana BioSciences
Locations (47):
- United States (30):
  - Pinnacle Research Group, LLC, Anniston, Alabama
  - Total Skin and Dermatology Center, PC., Birmingham, Alabama
  - Center for Dermatology Clinical Research, Inc., Fremont, California
  - L.A. Universal Research Center, Inc., Los Angeles, California
  - Dermatology Research Associates, Los Angeles, California
  - Revival Research, Doral, Florida
  - Clinical Physiology Associates, Fort Myers, Florida
  - Leavitt Medical Associates of Florida, Ormond Beach, Florida
  - Dermatology Consulting Services, Tampa, Florida
  - Forward Clinical Trials, Tampa, Florida
  - Dawes Fretzin Clinical Research Group, Indianapolis, Indiana
  - Dermatology Center of Indiana, PC, Plainfield, Indiana
  - The Indiana Clinical Trials Center, Plainfield, Indiana
  - Central Kentucky Research Associates, LLC, Lexington, Kentucky
  - Dermatology Specialists Research, Louisville, Kentucky
  - ActivMed Practices and Research, Inc., Portsmouth, New Hampshire
  - Corning Center for Clinical Research, Corning, New York
  - Mt. Sinai Hospital, New York, New York
  - Wake Research Associates, LLC, Raleigh, North Carolina
  - Dermatologists of Greater Colombus, Bexley, Ohio
  - Wright State Physicians, Fairborn, Ohio
  - Unity Clinical Research, Oklahoma City, Oklahoma
  - Vital Prospects Clinical Research Institute, Tulsa, Oklahoma
  - DermDox Centers for Dermatology, Hazleton, Pennsylvania
  - Synexus, Greer, South Carolina
  - Dermatology Treatment and Research Center, Dallas, Texas
  - Innovate Research, LLC, Fort Worth, Texas
  - The Center for Skin Research, Houston, Texas
  - Progressive Clinical Research, San Antonio, Texas
  - Virginia Clinical Research, Inc., Norfolk, Virginia
- Canada (7):
  - Institute of Skin Advancement Medical, Surgical, Costmetic & Laser Dermatology, Calgary
  - Innovaderm Research, Inc., Montreal
  - Ontario Inc., Ottawa
  - York Regional Dermatology, Richmond Hill
  - NewLab Clinical Research, Inc., St. John's
  - AvantDerm, Toronto
  - SkinWISE Dermatology, Winnipeg
- Germany (10):
  - Fachklinik Bad Bentheim, Bad Bentheim
  - Charité - Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Bonn AöR, Bonn
  - Universitätsklinikum Dresden, Dresden
  - Universitätsklinikum Frankfurt, Frankfurt
  - SRH Wald-Klinikum Gera GmbH, Gera
  - MENSINGDERMA research GmbH, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Schleswig-Holstein, Lübeck
  - Universitätshautklinik Münster, Münster

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Patient Enrolled July 5, 2018 Last Patient Out August 14, 2019
Period: Overall Study
Arm/Group | ASN002 40 mg | ASN002 60 mg | ASN002 80 mg | Placebo Oral Tablet
Started (Initially 62 subjects randomized into ASN002 40 mg arm, but one subject did not received any dose, therefore the subject was excluded from all analysis sets, including mITT and safety sets. The 10 subjects who were not completed the study in ASN002 40 mg group did not include the subjects who did not received any dose.) | 61 | 59 | 63 | 60
Completed | 51 | 54 | 49 | 49
Not Completed | 10 | 5 | 14 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ASN002 40 mg | ASN002 60 mg | ASN002 80 mg | Placebo Oral Tablet | Total
Number analyzed (Participants) | 61 | 59 | 63 | 60 | 243
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 57 | 50 | 56 | 56 | 219
  >=65 years | 4 | 9 | 7 | 4 | 24
Age, Continuous [Median (Full Range); unit: years] | 40 [18 to 71] | 36 [18 to 71] | 39 [19 to 75] | 42 [20 to 75] | 40 [18 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 28 | 32 | 31 | 125
  Male | 27 | 31 | 31 | 29 | 118
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 11 | 17 | 13 | 51
  Not Hispanic or Latino | 51 | 46 | 46 | 47 | 190
  Unknown or Not Reported | 0 | 2 | 0 | 0 | 2
Region of Enrollment [Number; unit: participants]
  Canada | 6 | 6 | 4 | 5 | 21
  United States | 47 | 43 | 51 | 47 | 188
  Germany | 8 | 10 | 8 | 8 | 34

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Eczema Area and Severity Index (EASI) at Week 12
Description: The Eczema Area and Severity Index (EASI) is a composite score ranging from 0 to 72, the higher the value the worse the disease, that takes into account the degree of erythema, induration/infiltration (papules), excoriation, and lichenification (each scored from 0 to 3 separately) for each of four body regions, with adjustment for the percentage of BSA involved for each body region and for the proportion of the body region to the whole body.
Time Frame: Week 12
Population: mITT
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ASN002 40 mg | ASN002 60 mg | ASN002 80 mg | Placebo Oral Tablet
Number analyzed (Participants) | 61 | 59 | 63 | 60
score on a scale | -15.8 (10.88) | -15.8 (9.82) | -17.5 (11.6) | -13.1 (11.87)

2. Secondary Outcome: Percent of Participant With at Least a 75% Reduction From Baseline in Eczema Area and Severity Index (EASI75)
Description: Percent of participants with at least a 75% reduction from baseline in EASI (EASI75) at Week 12
Time Frame: Week 12
Population: mITT (compared to PP all participants qualified for mITT were included but missing data were not imputed and not included in the percentages calculations)
Measure: Number; unit: percentage of patients
Arm/Group | ASN002 40 mg | ASN002 60 mg | ASN002 80 mg | Placebo Oral Tablet
Number analyzed (Participants) | 61 | 59 | 63 | 60
percentage of patients | 49 | 48.9 | 48.8 | 38.1

3. Secondary Outcome: Change From Baseline in 5-D Pruritus (Itching) Scale
Description: The 5-D Pruritus Scale is a 1-page, 5-question, validated questionnaire used in clinical trials to assess 5 dimensions of background itch: degree, duration, direction, disability, and distribution. Each question corresponds to 1 of the 5 dimensions of itch; subjects rated their symptoms over the preceding 2-week period as "present" or on a 1 to 5 scale, with 5 being the most affected. The total score of 5-D pruritus is a sum of the 5 scores to provide a total score range from 5 (best) to 25 (worst).
Time Frame: Week 12
Population: mITT (MMRM model was used)
Measure: Mean (Standard Deviation); unit: change in score on a scale
Arm/Group | ASN002 40 mg | ASN002 60 mg | ASN002 80 mg | Placebo Oral Tablet
Number analyzed (Participants) | 61 | 59 | 63 | 60
change in score on a scale | -6.6 (5.29) | -6.7 (4.48) | -6.3 (5.14) | -5.1 (4.47)

4. Secondary Outcome: Percent Change From Baseline in SCORing Atopic Dermatitis (SCORAD)
Description: In the SCORAD grading system, six items (erythema, edema/papulation, oozing/crusts, excoriation, lichenification, and dryness) evaluate the Atopic Dermatitis severity. The overall body surface area affected by atopic dermatitis was evaluated (from 0% to 100%) and included in the SCORAD scores. Loss of sleep and pruritus were evaluated by subjects on a visual analog scale (0-10) and were based on the average of the last three days/nights. The sum of these measures represented the SCORAD, which could range from 0 to 103. The higher the score the more severe the disease.
Time Frame: Week 12
Population: mITT (MMRM model was used to analyze the data)
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | ASN002 40 mg | ASN002 60 mg | ASN002 80 mg | Placebo Oral Tablet
Number analyzed (Participants) | 61 | 59 | 63 | 60
percentage change from baseline | -45.0 (33.81) | -47.3 (28.41) | -48.8 (28.02) | -38.5 (31.66)

5. Secondary Outcome: Percentage of Participants With a Response of Investigator's Global Assessment (IGA) 0 or 1
Description: The IGA is a global assessment of the current state of the disease. It is a 5-point (0-4) morphological assessment of overall disease severity. The 0 is the least severe and 4 is the most severe.
Time Frame: Week 12
Population: All patients with evaluable data at Week 12.
Measure: Number; unit: percentage of patients
Arm/Group | ASN002 40 mg | ASN002 60 mg | ASN002 80 mg | Placebo Oral Tablet
Number analyzed (Participants) | 49 | 47 | 43 | 42
percentage of patients | 26.5 | 29.8 | 23.3 | 19.0

6. Secondary Outcome: Change From Baseline in Patient-Oriented Eczema Measure (POEM)
Description: The Patient-Oriented Eczema Measure (POEM) is a self-assessment of disease severity by the subject. The POEM has a maximum value of 28 based on the subject's response to seven questions scored from 0 to 4. The higher the value the more severe the disease is.
Time Frame: Week 12
Population: Change from baseline at Week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ASN002 40 mg | ASN002 60 mg | ASN002 80 mg | Placebo Oral Tablet
Number analyzed (Participants) | 49 | 47 | 42 | 41
score on a scale | -8.9 (8.37) | -8.5 (8.1) | -9.1 (7.91) | -5.4 (6.47)

7. Secondary Outcome: Change From Baseline in Dermatology Life Quality Index (DLQI)
Description: Dermatology Life Quality Index Questionnaire (DLQI) is a simple 10-question validated questionnaire that has been used in more than 40 different skin conditions. The DLQI total score is defined as the sum of the 10 item scales, ranging from 0 to 30. The higher the value, the more severe the disease is.
Time Frame: Week 12
Population: All patients with available data at Week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ASN002 40 mg | ASN002 60 mg | ASN002 80 mg | Placebo Oral Tablet
Number analyzed (Participants) | 49 | 47 | 43 | 41
score on a scale | -8.1 (8.28) | -5.9 (6.59) | -8.5 (5.64) | -5.5 (6.48)

8. Secondary Outcome: Change From Baseline in Body Surface Area (BSA)
Description: The overall body surface area (BSA) affected by atopic dermatitis is evaluated (from 0% to 100%).
Time Frame: Week 12
Population: All patients with available data at Week 12
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | ASN002 40 mg | ASN002 60 mg | ASN002 80 mg | Placebo Oral Tablet
Number analyzed (Participants) | 49 | 47 | 43 | 42
percentage change from baseline | -57.2 (36.22) | -51.1 (51.6) | -50.1 (53.57) | -38.1 (47.65)

ADVERSE EVENTS:
Time Frame: 1 year, 1 month
Arm/Group | ASN002 40 mg | ASN002 60 mg | ASN002 80 mg | Placebo Oral Tablet
All-Cause Mortality (participants affected / at risk) | 0/61 | 0/59 | 0/63 | 0/60
Serious Adverse Events (participants affected / at risk) | 4/61 | 0/59 | 2/63 | 0/60
Other Adverse Events (participants affected / at risk) | 20/61 | 19/59 | 24/63 | 9/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ASN002 40 mg (N=61) | ASN002 60 mg (N=59) | ASN002 80 mg (N=63) | Placebo Oral Tablet (N=60)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
dysarthria (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
staphylococcal bacteremia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ASN002 40 mg (N=61) | ASN002 60 mg (N=59) | ASN002 80 mg (N=63) | Placebo Oral Tablet (N=60)
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 8 (8) | 4 (5) | 5 (5)
Headache (Nervous system disorders) | 6 (6) | 7 (7) | 4 (4) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (5) | 4 (4) | 5 (5) | 2 (2)
Urinary tract infection (Renal and urinary disorders) | 4 (4) | 0 (0) | 2 (2) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 6 (8) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 4 (5) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-02-07): https://cdn.clinicaltrials.gov/large-docs/57/NCT03531957/Prot_002.pdf
  • Statistical Analysis Plan (2019-08-12): https://cdn.clinicaltrials.gov/large-docs/57/NCT03531957/SAP_003.pdf